CLINICAL TRIAL: NCT01527266
Title: The Impact of a Sucrose Mouth-rinse in the Fasted and Fed-state on Time Trial Performance
Brief Title: Carbohydrate Mouth-rinse
Acronym: CHO rinse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 11-3-068
Record Dates: First submitted 2012-01-12; First posted 2012-02-06 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2012-10

CONDITIONS: Carbohydrate Mouth-rinse on Time Trial Performance
Keywords: carbohydrate; performance; cycling

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- carbohydrate mouth rinse fasted (Experimental): sucrose mouth rinse in the fasted state
  Interventions: Dietary Supplement: Carbohydrate drink
- carbohydrate mouth rinse fed (Experimental): sucrose mouth rinse fed state
  Interventions: Dietary Supplement: Carbohydrate drink
- Placebo mouth rinse fed (Placebo Comparator): placebo (non-caloric sweetened drink) in the fed state
  Interventions: Dietary Supplement: Placebo mouth rinse
- Placebo mouth rinse fasted (Placebo Comparator): placebo (non-caloric sweetened drink) in the fasted condition
  Interventions: Dietary Supplement: Placebo mouth rinse

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink — sucrose beverage
  Arms: carbohydrate mouth rinse fasted; carbohydrate mouth rinse fed
Dietary Supplement: Placebo mouth rinse — placebo; non-caloric sweetened beverage for use as a mouth rinse
  Arms: Placebo mouth rinse fasted; Placebo mouth rinse fed

SUMMARY:
Several studies have reported that carbohydrate (CHO) ingestion can improve performance during exercise of short duration (less than 60 min). However, there is no apparent metabolic explanation for this observation because endogenous CHO stores should not be a limiting factor during short duration exercise. Nonetheless, several groups have attempted to investigate CHO administration during short duration exercise with varying results. When CHO was administered intravenously, no performance effect was observed despite greater plasma glucose availability (5). Therefore, it was suggested that during exercise of short duration, exogenous CHO ingestion may exert its ergogenic effect by action through the central nervous system, possibly mediated by glucose receptors in the mouth. The latter has been investigated using a CHO-mouth rinse, whereby the CHO solution is spat out to remove any influence of the gut on exogenous CHO oxidation or performance. Using this rinse, studies have demonstrated results both for (5, 16), and against (1, 19) any improvement in short duration exercise performance when compared with a placebo. The discrepancy in the findings may be due to testing subjects in the fed (1) or fasted-state (5), when liver glycogen stores may be compromised. However, no study has tested subjects in both the fasted and fed-state using a CHO-mouth rinse. It remains to be determined whether CHO-mouth rinse is only effective at improving short duration exercise performance when subjects are in the fasted, compared with the fed-state. The investigators will test the hypothesis that CHO-mouth rinse improves performance in the fasted-state only compared with a placebo-rinse.

DETAILED DESCRIPTION:
It has been well established that carbohydrate (CHO) ingestion during prolonged, moderate- to high-intensity endurance-type exercise can delay the onset of fatigue and enhance exercise performance. Interestingly, several studies have reported that CHO ingestion can also improve performance during more intense exercise of short duration-less than 45-60 min. However, there is no apparent metabolic explanation for this improvement, because endogenous CHO stores should not limit exercise performance during short duration exercise tasks. To examine exogenous and endogenous glucose kinetics during high-intensity cycling exercise, Carter and colleagues tested 6 endurance athletes for 1 h at 75% Wmax while infusing either 20% glucose or 0.9% saline. Despite greater plasma glucose availability in the glucose-infusion trial, total CHO oxidation rates did not differ between treatments. Moreover, no performance benefits were observed after intravenous glucose administration. Consequently, the authors suggested that CHO ingestion during high-intensity exercise of short duration might exert its ergogenic effect by acting through the central nervous system, possibly mediated by glucose receptors in the mouth or gastrointestinal tract.

To test this hypothesis, Carter and colleagues investigated the impact of a carbohydrate mouth-rinse solution on 1-h time trial performance. The use of a mouth-rinse treatment, in which a CHO solution is spat out without swallowing, was chosen to remove any influence of the gut or exogenous CHO oxidation on performance. Participants were reported to cycle faster after a mouth rinse with a 6.4% maltodextrin solution at every 12.5% of the trial completed compared with a placebo rinse. The authors concluded that CHO mouth rinsing improves time trial performance and that the mechanism responsible might be an increase in central drive or motivation mediated by glucose receptors in the mouth. However in the former study, subjects were tested in a fasted state, which is impractical compared to how athletes normally prepare for training and competition.

In follow-up to the former study, we tested the performance effect of a carbohydrate mouth rinse 2 h after subjects ingested a CHO rich meal. From an evolutionary viewpoint, it can be speculated that the potential stimulating effect of glucose in the mouth might be of considerable impact under conditions when liver glycogen stores might be compromised. In agreement with this theory, there was no performance improvement with a CHO mouth rinse during time trial performance 2 h following the ingestion of a CHO -rich meal. However, as there are now studies demonstrating results both for and against any ergogenic effect of a CHO mouth rinse during short duration time trials it remains to be determined whether CHO mouth rinse improves performance during a 1 h time trial in the fasted state only. Therefore, the present study aims to investigate any potential ergogenic effect of a CHO mouth rinse during a 1 h time trial performance in both the fasted and fed state.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* 18 - 35 years of age
* Endurance cycling trained (≥ 3 sessions of endurance exercise per week)
* VO2 max ≥ 50 ml/kg/min
* Training history of more than one year of ≥ 3 sessions of endurance cycling exercise per week
* BMI < 25 kg/m2

Exclusion Criteria:

* Use of medication
* Smoking

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Time to complete a set amount of work (time-trial performance) | laboratory visit 2
  Time to complete the set amount of work measured in minutes. To determine if one intervention allows the subject to complete the given amount of work in a faster time period than the placebo.
Time to complete a set amount of work (time trial performance) | laboratory visit 3
  Time to complete the set amount of work measured in minutes. To determine if one intervention allows the subject to complete the given amount of work in a faster time period than the placebo.
Time to complete a set amount of work (time-trial performance) | laboratory visit 4
  Time to complete the set amount of work measured in minutes. To determine if one intervention allows the subject to complete the given amount of work in a faster time period than the placebo.
Time to complete a set amount of work (time-trial performance) | laboratory visit 5
  Time to complete the set amount of work measured in minutes. To determine if one intervention allows the subject to complete the given amount of work in a faster time period than the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Luc van Loon, Ph.D., Study Director — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Netherlands